CLINICAL TRIAL: NCT02580981
Title: Acute Lymphoblastic Leukemia Therapies Informed by Genomic Analyses
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Staffing
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INST UNM 1503
Record Dates: First submitted 2015-10-05; First posted 2015-10-20 (Estimated); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Leukemia, Acute Lymphoblastic
Keywords: Cancer; Oncology; Acute Lymphoblastic Leukemia; ALL; Genomics; Genetics; Sequencing; DNA; RNA; Ph-like
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Genomic Testing (Experimental): Newly diagnosed ALL patients will undergo genomic studies listed in Primary Objective 1. Analyses will be performed on a bone marrow (BM) aspirate at initial diagnosis (patients with an absolute blast count of at least 1,000/μL, may submit 2 mL of peripheral blood at diagnosis for each 1 mL of required BM. In patients in whom the aspirate cannot be obtained, a core biopsy will be used).
  In addition, flow cytometric analysis and deep sequencing will be used to characterize and monitor the molecular heterogeneity and clonal evolution of disease during front-line therapy. BM, blood, and buccal specimens will be collected on day 29 of induction treatment and possibly at a later time point if relapse occurs.
  Interventions: Other: Acute Lymphobastic Leukemia (ALL) Treatment Options

INTERVENTIONS:
Other: Acute Lymphobastic Leukemia (ALL) Treatment Options — Depending on the genomic testing results, patients with targetable genomic lesions will be enrolled onto available national clinical trials that are sponsored by the NCI National Clinical Trials Network (NCTN) (COG and other adult NCI Cooperative Groups). If no suitable NCTN trial exists, appropriate therapeutic regimens (including currently accepted standards-of-care), alterations in therapy, or treatment with targeted agents to specific genomic lesions will be considered.

SUMMARY:
Previous work performed by University of New Mexico Comprehensive Cancer Center (UNMCCC) investigators has revealed previously unknown genomic mutations in children, adolescents, and young adults with high-risk B and T cell precursor acute lymphoblastic leukemia (ALL). Using genomic and next generation DNA sequencing technologies, these investigators revealed that 14% of children with high-risk ALL have "Philadelphia chromosome-like" ("Ph-like") ALL. Patients with this form of ALL were found to have a significantly increased risk of treatment failure and death.

Further work revealed that there are more than 40 distinct gene rearrangements and fusions that can result in Ph-like ALL. Cell lines and human leukemic cells expressing some of these different gene fusions were sensitive to currently available drugs. This suggests that Ph-like ALL patients with these specific distinct gene fusions should be targeted in future clinical trials to be treated with appropriate therapy. Further work is also needed to identify other potentially targetable genetic alterations in ALL patients.

Therefore, the goal of this study is to perform genomic screening of all newly diagnosed ALL patients seen at UNM and to use this information to enroll patients onto available National Clinical Trial Network (NCTN) clinical trials. If an appropriate NCTN trial is not available, best clinical management will be pursued.

DETAILED DESCRIPTION:
The work performed by UNMCCC investigators and others as described briefly above has provided major insights into the biologic and clinical features and the genomic landscape of Ph-like ALL, which is strikingly heterogeneous. Gene expression profiling and RNA/transcriptomic, exome, and whole genome sequencing have identified several distinct subclasses of kinase activating lesions in 91% of the Ph-like ALL cases studied to date, most commonly kinase and cytokine receptor gene rearrangements and fusions. UNMCCC investigators are now collaborating with Children's Oncology Group (COG) and the adult National Cancer Institute (NCI) Cooperative Groups (Southwest Oncology Group (SWOG), Eastern Cooperative Oncology Group (ECOG) - American College of Radiology Imaging Network (ACRIN), The Alliance) to develop national clinical trials for pediatric, adolescent and young adult (AYA), and adult ALL patients that incorporate their genomic diagnostic screens, molecular diagnostics, and next generation sequencing studies to identify underlying genomic lesions in ALL and target patients to appropriate therapeutic regimens.

In this feasibility study, next generation sequencing (NGS) technologies will inform an acute lymphoblastic leukemia risk classification system, which may be adapted to identify patients who might benefit from targeted therapies; such patients will be targeted to NCTN National Treatment trials or UNMCCC-sponsored trials where appropriate, through detailed genomic data analysis performed under College of American Pathologists (CAP)/CLIA conditions and in individual case discussions in a Molecular Tumor Board.

In addition, the association of race and ethnicity with the spectrum of ALL-associated genomic mutations in the New Mexico and regional ALL population, which includes a significant proportion of underrepresented minorities, will be studied. This may ultimately allow for the development of an ancestry-based risk classification system.

ELIGIBILITY:
Inclusion Criteria:

* New diagnosis of Acute Lymphoblastic Leukemia
* No previous therapy, excluding emergency radiation, steroids or intrathecal cytarabine
* Any age
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Previous therapy, excluding emergency radiation, steroids or intrathecal cytarabine
* Not willing to obtain cancer care at the University of New Mexico

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-07-28 (Actual); Primary Completion 2022-03-19 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
ALL characterization: Low Density Array | 3 years
  Newly diagnosed ALL patients at UNMCCC will undergo Low Density Array (LDA) card screening (a gene expression classifier for Ph-like ALL) at initial diagnosis. The proportion of LDA status (positive vs. negative) and its 95% confidence interval will be calculated based on the exact binomial distribution.
ALL characterization: Next Generation Sequencing | 3 years
  Newly diagnosed ALL patients at UNMCCC will undergo Next Generation Sequencing (NGS) at initial diagnosis. NGS (exomic and transcriptomic) of a sufficient read depth (500-700x) will be employed to detect clonal heterogeneity at diagnosis. Statistical analysis will be primarily descriptive (e.g. frequency (proportion) of various mutations will be calculated).
ALL characterization: SNP analysis | 3 years
  Newly diagnosed ALL patients at UNMCCC will undergo Molecular Determination of Genetic Ancestry (using a panel of single nucleotide polymorphisms (SNPs)) at initial diagnosis. Statistical analysis will be primarily descriptive (e.g. frequency (proportion) of SNPs and genetic ancestry groups will be calculated)

SECONDARY OUTCOMES:
Relationship of patient characteristics to trial enrollment | 3 years
  Genetic and molecular characterization as described for the Primary Outcome Measures will be summarized for patients who are enrolled on NCTN clinical trials and for those who are not enrolled on NCTN clinical trials. The two group comparisons (NCTN vs. non-NCTN) will be tested using non-parametric approach such as Wilcoxon sum rank test.
Relationship between race/ethnicity and outcome | 3 years
  Time-to-event data (such as Progression free survival (PFS), determined clinically) will be summarized using Kaplan-Meier curves along with log-rank test by the treatment groups as well as race/ethnicity determined through molecular assessment of genetic ancestry as described in Primary Outcome Measure 3. Multivariable Cox Proportional Hazards model will also be explored for PFS with treatment and/or ethnicity variables.
Feasibility of discovering molecular features in ALL with therapeutic relevance | 3 years
  Feasibility will be assessed by calculation of the following statistics: percent of patients who enrolled in NCTN trials, percent of patients with minimal residual disease (MRD) that are completely evaluated over time, percent of patients for whom molecularly characterization is feasible and informative over the treatment course. All estimated proportions will be accompanied by exact 95% confidence intervals
Minimal Residual Disease (MRD) evaluation | 3 years
  End-induction Minimal Residual Disease (MRD) will be performed using a Clinical Laboratory Improvement Amendments (CLIA)-approved flow-cytometric assay at the Children's Oncology Group University of Washington Reference Laboratory. Molecular MRD will also be determined using research-based deep sequencing. MRD repeatedly measured across time points will be summarized using descriptive statistics (bar graph for High vs. Low status). Associations between the MRD and the treatment groups (LAD Positive vs. LAD Negative for NCTN and Non-NCTN treatment groups), using the exact Pearson Chi-Square test with Monte Carlo simulation at each time point will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Jodi Mayfield, MD, Principal Investigator — University of New Mexico, Department of Pediatrics
Locations (1):
- University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of New Mexico Comprehensive Cancer Center — http://www.cancer.unm.edu
- See also: New Mexico Cancer Care Alliance — http://www.nmcca.org